CLINICAL TRIAL: NCT00319098
Title: A Phase III, Observer-blind, Randomised Study to Evaluate the Safety and Immunogenicity of One and Two Administrations of Pandemic Monovalent (H5N1) Influenza Vaccine (Adjuvanted Split Virus Formulation) in Adults Aged 18 Years and Older
Brief Title: Study to Evaluate the Safety and Immunogenicity of a Pandemic Influenza Vaccine in Adults Aged 18 Years and Above
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 107064; 107217 (Other: GSK)
Record Dates: First submitted 2006-04-26; First posted 2006-04-27 (Estimated); Results first posted 2017-08-03 (Actual); Last update posted 2018-07-23 (Actual); Status verified 2017-04

CONDITIONS: Influenza
Keywords: Adjuvanted pandemic influenza candidate vaccine; Influenza
MeSH Terms: conditions — Influenza, Human | interventions — fluarix

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- GSK1562902A Group (Experimental): Male and female subjects aged 18 or over received two intramuscular doses of the GSK1562902A study vaccine, at Day 0 and Day 21, into the non-dominant arm. The group was further stratified by age for analyses.
  Interventions: Biological: Adjuvanted pandemic influenza candidate vaccine
- Fluarix+Placebo Group (Active Comparator): Male and female subjects aged 18 or over received one dose of Fluarix™ vaccine at Day 0 and one dose of placebo at Day 21, intramuscularly into de non-dominant arm. The group was further stratified by age for analyses.
  Interventions: Biological: Fluarix; Biological: Placebo

INTERVENTIONS:
Biological: Adjuvanted pandemic influenza candidate vaccine — 2 doses, intramuscular injection
  Arms: GSK1562902A Group
Biological: Fluarix — One intramuscular injection
  Arms: Fluarix+Placebo Group
Biological: Placebo — One intramuscular injection
  Arms: Fluarix+Placebo Group

SUMMARY:
Today, the leading contender for the next pandemic of influenza is H5N1, a strain of avian virus. Prevention and control will depend on the rapid production and worldwide distribution of specific pandemic vaccines. Candidate 'pandemic-like' vaccines must be developed and tested in clinical trials to determine the most optimal formulation and the best vaccination schedule. This study is designed to test in healthy adults aged above 18 years the reactogenicity and immunogenicity of one and two administrations of a candidate pandemic H5N1 vaccine formulated from Split Virus.

DETAILED DESCRIPTION:
This study has 2 phases:

The study ID 107064 corresponds to objectives & outcome measures evaluated from day 0 until day 51.

The study ID 107217 corresponds to objectives & outcome measures evaluated at day 180.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol.
* A male or female aged 18 years or above at the time of the first vaccination.
* Written informed consent obtained from the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* If the subject is female, she must be of non-childbearing potential, for 30 days prior to first vaccination, have a negative pregnancy test and must agree to continue such precautions for two months after completion of the vaccination series.

Exclusion Criteria:

* Administration of other licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to enrolment in this study. Planned administration of a vaccine not foreseen by the study protocol up to 30 days after the second vaccination.
* Administration of interpandemic influenza vaccine between Day 0 and Day 51of the study. Those study participants belonging to risk groups eligible to receive the annual interpandemic influenza vaccine (in accordance with local regulations) can receive the annual vaccination after day 51 and before the end of the study on Day 180.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within 6 months prior to the first administration of the study vaccine.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination
* History of chronic alcohol consumption and/or drug abuse.
* History of hypersensitivity to vaccines.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Acute clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Major congenital defects or serious chronic disease including any medically significant chronic pulmonary, cardiovascular, renal, neurological, psychiatric or metabolic disorder, as determined by medical history and physical examination. (Subjects suffering from seasonal allergies or asthma under inhalative treatment can be included).
* Acute disease at the time of enrolment.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the first administration of the study vaccine or during the study.
* Lactating women
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days prior to the first vaccination, or planned use during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5075 (Actual)
Dates: Start 2006-05-01 (Actual); Primary Completion 2007-01-01 (Actual); Study Completion 2007-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (29):
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- France (6):
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Lagord
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Poitiers
  - GSK Investigational Site, Rouen
- Germany (10):
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Regensburg, Bavaria
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Schwerin, Mecklenburg-Vorpommern
  - GSK Investigational Site, Witten, North Rhine-Westphalia
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- GSK Investigational Site, Rotterdam, Netherlands
- Russia (4):
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Novokuznetsk
  - GSK Investigational Site, Saratov
  - GSK Investigational Site, Yekaterinburg
- Spain (4):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Marid
  - GSK Investigational Site, Valencia
- Sweden (2):
  - GSK Investigational Site, Eskilstuna
  - GSK Investigational Site, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Rumke HC, Bayas JM, de Juanes JR, Caso C, Richardus JH, Campins M, Rombo L, Duval X, Romanenko V, Schwarz TF, Fassakhov R, Abad-Santos F, von Sonnenburg F, Drame M, Sanger R, Ballou WR. Safety and reactogenicity profile of an adjuvanted H5N1 pandemic candidate vaccine in adults within a phase III safety trial. Vaccine. 2008 May 2;26(19):2378-88. doi: 10.1016/j.vaccine.2008.02.068. Epub 2008 Mar 27. PMID 18407382
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 107064 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 107064 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 107064 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 107064 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 107064 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register. The results of this study 107064 are summarised with study 107217 on the GSK Clinical Study Register.
- Available data/document: Statistical Analysis Plan: 107064 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of the 5075 subjects enrolled in this study, 4 subjects did not receive any study vaccine and were hence excluded from study start.
Period: Overall Study
Arm/Group | GSK1562902A Group | Fluarix+Placebo Group
Started | 3802 | 1269
Completed | 3667 | 1237
Not Completed | 135 | 32
Not completed — Serious adverse event | 3 | 0
Not completed — Adverse Event | 20 | 1
Not completed — Withdrawal by Subject | 37 | 8
Not completed — Migrated/moved from study area | 2 | 1
Not completed — Lost to Follow-up | 37 | 13
Not completed — Others | 33 | 8
Not completed — Protocol Violation | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- GSK1562902A 18-60 YOA Group: Male and female subjects 18-60 years of age (YOA) received two intramuscular doses of the GSK1562902A study vaccine, at Day 0 and Day 21, into the non-dominant arm.
- GSK1562902A >60 YOA Group: Male and female subjects over (>) 60 years of age (YOA) received two intramuscular doses of the GSK1562902A study vaccine, at Day 0 and Day 21, into the non-dominant arm.
- Fluarix+Placebo 18-60 YOA Group: Male and female subjects 18-60 years of age (YOA) received one dose of Fluarix™ vaccine at Day 0 and one dose of placebo at Day 21, intramuscularly into de non-dominant arm.
- Fluarix+Placebo >60 YOA Group: Male and female subjects over (>) 60 years of age (YOA) received one dose of Fluarix™ vaccine at Day 0 and one dose of placebo at Day 21, intramuscularly into de non-dominant arm.
- Total: Total of all reporting groups
Arm/Group | GSK1562902A 18-60 YOA Group | GSK1562902A >60 YOA Group | Fluarix+Placebo 18-60 YOA Group | Fluarix+Placebo >60 YOA Group | Total
Number analyzed (Participants) | 3397 | 405 | 1136 | 133 | 5071
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.8 (12.24) | 67.3 (6.01) | 35.4 (12.51) | 66.6 (5.20) | 38.36 (15.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2018 | 187 | 691 | 56 | 2952
  Male | 1379 | 218 | 445 | 77 | 2119

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Solicited Local Symptoms
Description: Assessed solicited local symptoms were ecchymosis, induration, pain, redness and swelling. Any = occurrence of symptom regardless of intensity grade. Grade 3 Pain = pain that prevented normal everyday activities Grade 3 ecchymosis/induration/redness/swelling = redness/swelling spreading beyond (>) 50 millimeters (mm) in diameter
Time Frame: During a 7 day follow-up period after each dose of vaccine and overall.
Population: The analysis was performed on the Total Vaccinated cohort (TVc) which included all vaccinated subjects for whom data were available and with the symptom sheet filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A 18-60 YOA Group | GSK1562902A >60 YOA Group | Fluarix+Placebo 18-60 YOA Group | Fluarix+Placebo >60 YOA Group
Number analyzed (Participants) | 3343 | 403 | 1123 | 133
Participants
  Any Ecchymosis, Dose 1 [N=3342;403;1123;133] | 212 | 16 | 39 | 3
  Grade 3 Ecchymosis, Dose 1[N=3342;403;1123;133] | 8 | 1 | 0 | 0
  Any Induration, Dose 1[N=3342;403;1123;133] | 876 | 73 | 199 | 17
  Grade 3 Induration, Dose 1[N=3342;403;1123;133] | 96 | 6 | 10 | 0
  Any Pain, Dose 1[N=3342;403;1123;133] | 2926 | 233 | 724 | 36
  Grade 3 Pain, Dose 1[N=3342;403;1123;133] | 169 | 3 | 6 | 0
  Any Redness, Dose 1[N=3342;403;1123;133] | 910 | 112 | 281 | 34
  Grade 3 Redness, Dose 1[N=3342;403;1123;133] | 128 | 12 | 17 | 0
  Any Swelling, Dose 1[N=3342;403;1123;133] | 812 | 88 | 176 | 15
  Grade 3 Swelling, Dose 1[N=3342;403;1123;133] | 134 | 12 | 12 | 1
  Any Ecchymosis, Dose 2 [N=3247;395;1102;132] | 144 | 16 | 31 | 3
  Grade 3 Ecchymosis, Dose 2 [N=3247;395;1102;132] | 3 | 1 | 1 | 0
  Any Induration, Dose 2 [N=3247;395;1102;132] | 734 | 75 | 41 | 5
  Grade 3 Induration, Dose 2 [N=3247;395;1102;132] | 81 | 7 | 0 | 0
  Any Pain, Dose 2 [N=3247;395;1102;132] | 2451 | 199 | 173 | 8
  Grade 3 Pain, Dose 2 [N=3247;395;1102;132] | 77 | 1 | 2 | 0
  Any Redness, Dose 2 [N=3247;395;1102;132] | 819 | 105 | 93 | 16
  Grade 3 Redness, Dose 2 [N=3247;395;1102;132] | 168 | 25 | 1 | 0
  Any Swelling, Dose 2 [N=3247;395;1102.132] | 719 | 89 | 42 | 4
  Grade 3 Swelling, Dose 2 [N=3247;395;1102;132] | 96 | 11 | 0 | 0
  Any Ecchymosis, Across [N=3343;403;1123;133] | 320 | 29 | 65 | 5
  Grade 3 Ecchymosis, Across [N=3343;403;1123;133] | 11 | 2 | 1 | 0
  Any Induration, Across [N=3343;403;1123;133] | 1150 | 108 | 215 | 19
  Grade 3 Induration, Across [N=3343;403;1123;133] | 148 | 12 | 10 | 0
  Any Pain, Across [N=3343;403;1123;133] | 3037 | 271 | 748 | 39
  Grade 3 Pain, Across [N=3343;403;1123;133] | 221 | 4 | 8 | 0
  Any Redness, Across [N=3343;403;1123;133] | 1277 | 165 | 312 | 38
  Grade 3 Redness, Across [N=3343;403;1123;133] | 250 | 36 | 17 | 0
  Any Swelling, Across [N=3343;1123;133] | 1107 | 133 | 196 | 17
  Grade 3 Swelling, Across [N=3343;1123;133] | 189 | 22 | 12 | 1

2. Primary Outcome: Number of Subjects With Solicited General Symptoms (Dose 1)
Description: Assessed solicited general symptoms were arthralgia, fatigue, fever [defined as axillary temperature equal to or above (≥) 37.5 degrees Celsius (°C)], headache, myalgia, shivering, sweating. Any = occurrence of symptom regardless of intensity grade and relationship to vaccination. Grade 3 symptom = symptoms that prevented normal activity. Grade 3 Fever = fever higher than (>) 39.0 °C. Related = symptom considered by the investigator to be casually related with the study vaccination.
Time Frame: During the 7-day (Days 0-6) after Dose 1
Population: The analysis was performed on the TVc which included all vaccinated subjects for whom data were available and with the symptom sheet filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A 18-60 YOA Group | GSK1562902A >60 YOA Group | Fluarix+Placebo 18-60 YOA Group | Fluarix+Placebo >60 YOA Group
Number analyzed (Participants) | 3341 | 403 | 1123 | 133
Participants
  Any Arthralgia, Dose 1 | 625 | 57 | 100 | 13
  Grade 3 Arthralgia, Dose 1 | 47 | 1 | 3 | 1
  Related Arthralgia, Dose 1 | 583 | 46 | 86 | 11
  Any Fatigue, Dose 1 | 1384 | 80 | 284 | 20
  Grade 3 Fatigue, Dose 1 | 90 | 3 | 4 | 2
  Related Fatigue, Dose 1 | 1220 | 67 | 235 | 15
  Any Fever, Dose 1 | 270 | 10 | 24 | 6
  Grade 3 Fever, Dose 1 | 7 | 0 | 0 | 0
  Related Fever, Dose 1 | 243 | 8 | 20 | 5
  Any Headache, Dose 1 | 1159 | 79 | 275 | 18
  Grade 3 Headache, Dose 1 | 60 | 1 | 6 | 2
  Related Headache, Dose 1 | 960 | 63 | 203 | 15
  Any Myalgia, Dose 1 | 1336 | 93 | 239 | 12
  Grade 3 Myalgia, Dose 1 | 77 | 1 | 5 | 2
  Related Myalgia, Dose 1 | 1249 | 80 | 220 | 11
  Any Shivering, Dose 1 | 482 | 14 | 67 | 3
  Grade 3 Shivering, Dose 1 | 34 | 0 | 2 | 0
  Related Shivering, Dose 1 | 448 | 11 | 55 | 3
  Any Sweating, Dose 1 | 481 | 38 | 95 | 17
  Grade 3 Sweating, Dose 1 | 17 | 3 | 1 | 1
  Related Sweating, Dose 1 | 415 | 31 | 71 | 15

3. Primary Outcome: Number of Subjects With Solicited General Symptoms (Dose 2)
Description: as for outcome 2
Time Frame: During the 7-day (Days 0-6) after Dose 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A 18-60 YOA Group | GSK1562902A >60 YOA Group | Fluarix+Placebo 18-60 YOA Group | Fluarix+Placebo >60 YOA Group
Number analyzed (Participants) | 3246 | 395 | 1102 | 132
Participants
  Any Arthralgia, Dose 2 | 513 | 47 | 41 | 6
  Grade 3 Arthralgia, Dose 2 | 46 | 3 | 2 | 0
  Related Arthralgia, Dose 2 | 493 | 39 | 34 | 4
  Any Fatigue, Dose 2 | 1108 | 77 | 148 | 14
  Grade 3 Fatigue, Dose 2 | 81 | 2 | 5 | 1
  Related Fatigue, Dose 2 | 1014 | 66 | 119 | 12
  Any Fever, Dose 2 | 278 | 16 | 15 | 5
  Grade 3 Fever, Dose 2 | 10 | 1 | 0 | 0
  Related Fever, Dose 2 | 266 | 14 | 10 | 4
  Any Headache, Dose 2 | 934 | 69 | 155 | 8
  Grade 3 Headache, Dose 2 | 59 | 2 | 8 | 0
  Related Headache, Dose 2 | 800 | 56 | 111 | 8
  Any Myalgia, Dose 2 | 1044 | 72 | 67 | 10
  Grade 3 Myalgia, Dose 2 | 61 | 4 | 5 | 0
  Related Myalgia, Dose 2 | 999 | 65 | 53 | 7
  Any Shivering, Dose 2 | 390 | 15 | 24 | 5
  Grade 3 Shivering, Dose 2 | 29 | 1 | 0 | 0
  Related Shivering, Dose 2 | 378 | 13 | 19 | 5
  Any Sweating, Dose 2 | 442 | 41 | 59 | 13
  Grade 3 Sweating, Dose 2 | 32 | 7 | 2 | 1
  Related Sweating, Dose 2 | 397 | 33 | 42 | 9

4. Primary Outcome: Number of Subjects With Solicited General Symptoms (Across Doses)
Description: as for outcome 2
Time Frame: During the 7-day (Days 0-6) post vaccination across dosses
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A 18-60 YOA Group | GSK1562902A >60 YOA Group | Fluarix+Placebo 18-60 YOA Group | Fluarix+Placebo >60 YOA Group
Number analyzed (Participants) | 3342 | 403 | 1123 | 133
Participants
  Any Arthralgia, Across | 874 | 82 | 130 | 15
  Grade 3 Arthralgia, Across | 87 | 4 | 4 | 1
  Related Arthralgia, Across | 829 | 67 | 112 | 13
  Any Fatigue, Across | 1736 | 117 | 346 | 24
  Grade 3 Fatigue, Across | 155 | 4 | 8 | 3
  Related Fatigue, Across | 1576 | 100 | 289 | 17
  Any Fever, Across | 466 | 24 | 38 | 9
  Grade 3 Fever, Across | 16 | 1 | 0 | 0
  Related Fever, Across | 432 | 20 | 29 | 7
  Any Headache, Across | 1566 | 114 | 350 | 19
  Grade 3 Headache, Across | 112 | 3 | 14 | 2
  Related Headache, Across | 1347 | 94 | 266 | 16
  Any Myalgia, Across | 1670 | 124 | 276 | 18
  Grade 3 Myalgia, Across | 125 | 5 | 9 | 2
  Related Myalgia, Across | 1593 | 107 | 249 | 14
  Any Shivering, Across | 711 | 26 | 86 | 5
  Grade 3 Shivering, Across | 56 | 1 | 2 | 0
  Related Shivering, Across | 675 | 21 | 71 | 5
  Any Sweating, Across | 727 | 64 | 134 | 19
  Grade 3 Sweating, Across | 47 | 9 | 3 | 2
  Related Sweating, Across | 649 | 53 | 102 | 16

5. Primary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination. Related symptoms were not available.
Time Frame: During the 21st Day (Days 0-20) post Dose 1
Population: The analysis was performed on the TVc which included all vaccinated subjects for whom data were available and with the symptom sheet filled in at Day 51.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A 18-60 YOA Group | GSK1562902A >60 YOA Group | Fluarix+Placebo 18-60 YOA Group | Fluarix+Placebo >60 YOA Group
Number analyzed (Participants) | 3397 | 405 | 1136 | 133
Participants
  Any AEs | 917 | 74 | 244 | 19
  Grade 3 AEs | 95 | 5 | 22 | 1

6. Primary Outcome: Number of Subjects With AEs
Description: as for outcome 5
Time Frame: During the 30 Day (Days 0-29) post Dose 2
Population: The analysis was performed on the TVc which included all subjects who had received the second dose and for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A 18-60 YOA Group | GSK1562902A >60 YOA Group | Fluarix+Placebo 18-60 YOA Group | Fluarix+Placebo >60 YOA Group
Number analyzed (Participants) | 3267 | 396 | 1111 | 133
Participants
  Any AEs | 644 | 75 | 180 | 23
  Grade 3 AEs | 65 | 9 | 28 | 3

7. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: From Day 0 to Day 180
Population: The analysis was performed on the Vaccinated Cohort (Extended follow-up) which included all vaccinated subjects for whom data were available at Day 180.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A 18-60 YOA Group | GSK1562902A >60 YOA Group | Fluarix+Placebo 18-60 YOA Group | Fluarix+Placebo >60 YOA Group
Number analyzed (Participants) | 3253 | 390 | 1102 | 129
Participants | 27 | 15 | 10 | 5

8. Primary Outcome: Number of Subjects With New Onset Chronic Diseases (NOCDs)
Description: NOCDs include autoimmune disorders, asthma, type I diabetes, allergies.
Time Frame: From Day 0 to Day 180
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A 18-60 YOA Group | GSK1562902A >60 YOA Group | Fluarix+Placebo 18-60 YOA Group | Fluarix+Placebo >60 YOA Group
Number analyzed (Participants) | 3253 | 390 | 1102 | 129
Participants | 9 | 7 | 3 | 0

9. Primary Outcome: Number of Subjects With Medically Significant Conditions (MSCs)
Description: MSCs prompting emergency room or physician visits that were not related to common diseases or routine visits. Common diseases included upper respiratory infections, sinusitis, pharyngitis, gastroenteritis, urinary tract infections, cervico-vaginal yeast infections, menstrual cycle abnormalities and injury.
Time Frame: From Day 0 to Day 51
Population: The analysis was performed on the TVc which included all vaccinated subjects for whom data were available at Day 51.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A 18-60 YOA Group | GSK1562902A >60 YOA Group | Fluarix+Placebo 18-60 YOA Group | Fluarix+Placebo >60 YOA Group
Number analyzed (Participants) | 3397 | 405 | 1136 | 133
Participants | 60 | 10 | 11 | 3

10. Secondary Outcome: Anti- Haemagglutinin Antibody (Anti-HA) Titers Against Avian Influenza A Subtype H5N1
Description: Anti-HA antibody titers were expressed as Geometric Mean Tiyers (GMTs).
Time Frame: At Day 0 (PRE), 21 and 42
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity which included all evaluable subjects of the immunogenicity subset for whom data concerning immunogenicity endpoint measures were available. This includes subjects for whom assay results were available after vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK1562902A 18-60 YOA Group | GSK1562902A >60 YOA Group | Fluarix+Placebo 18-60 YOA Group | Fluarix+Placebo >60 YOA Group
Number analyzed (Participants) | 269 | 146 | 97 | 50
Titers
  anti-HA, Pre [N=269;146;96;50] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0]
  anti-HA, Day 21 [N=269;145;97;49] | 31.8 [25.7 to 39.4] | 43.8 [33.3 to 57.5] | 6.0 [5.1 to 7.0] | 7.5 [5.5 to 10.4]
  anti-HA, Day 42 [N=268;140;96;50] | 307.0 [258.4 to 364.8] | 187.0 [148.8 to 235.1] | 5.6 [4.9 to 6.3] | 7.5 [5.5 to 10.2]

11. Secondary Outcome: Number of Seroconverted Subjects Against H5N1
Description: Seroconversion rate for Haemagglutinin antibody response was defined as the number of vaccinees who had either a pre-vaccination titer lower than (<) 1:10 and a post-vaccination titer greater than or equal to (≥) 1:40 or a pre-vaccination titer ≥ 1:10 and at least a fourfold increase in post-vaccination titer. Seroconversion rate for Neutralising antibody response was defined as the percentage of vaccinees with a minimum 4-fold increase in titer at post-vaccination.
Time Frame: At Day 21 and Day 42
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A 18-60 YOA Group | GSK1562902A >60 YOA Group | Fluarix+Placebo 18-60 YOA Group | Fluarix+Placebo >60 YOA Group
Number analyzed (Participants) | 269 | 146 | 96 | 50
Participants
  anti-HA, Day 21 [N=269;145;96;49] | 147 | 89 | 5 | 5
  anti-HA, Day 42 [N=268;140;96;50] | 245 | 128 | 3 | 6

12. Secondary Outcome: Seroconversion Factor for Hemagglutination Inhibition (HI) Antibodies Against A/Vietnam Influenza Strain
Description: Seroconversion factor was defined as the fold increase in serum HI GMTs post-vaccination compared to day 0.
Time Frame: At Day 21 and Day 42
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: Titer fold increase
Arm/Group | GSK1562902A 18-60 YOA Group | GSK1562902A >60 YOA Group | Fluarix+Placebo 18-60 YOA Group | Fluarix+Placebo >60 YOA Group
Number analyzed (Participants) | 269 | 145 | 96 | 50
Titer fold increase
  A/Vietnam, Day 21 [N=269;145;96;49] | 6.4 [5.1 to 7.9] | 8.8 [6.7 to 11.5] | 1.2 [1.0 to 1.4] | 1.5 [1.1 to 2.1]
  A/Vietnam, Day 21 [N=268;140;96;50] | 61.4 [51.7 to 73.0] | 37.4 [29.8 to 47.0] | 1.1 [1.0 to 1.3] | 1.5 [1.1 to 2.0]

13. Secondary Outcome: Number of Seroprotected Subjects Against A/Vietnam Influenza Strain
Description: Seroprotection rate was defined as the number of vaccinees with a serum HI titer ≥1:40 that usually is accepted as indicating protection.
Time Frame: At Day 0 (PRE), Day 21 and Day 42
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A 18-60 YOA Group | GSK1562902A >60 YOA Group | Fluarix+Placebo 18-60 YOA Group | Fluarix+Placebo >60 YOA Group
Number analyzed (Participants) | 269 | 146 | 97 | 50
Participants
  A/Vietnam, PRE [N=269;146;96;50] | 0 | 0 | 0 | 0
  A/Vietnam, Day 21 [N=269;145;97;49] | 147 | 89 | 5 | 5
  A/Vietnam, Day 42 [N=268;140;96;50] | 245 | 128 | 3 | 6

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms during the 7 days post-vaccination, Unsolicited AEs during the 21 post Dose 1 and 30 days post Dose 2; SAEs from Day 0 to Day 180.
Description: During the given time frame for unsolicited AEs, no symptom reached nor surpassed the 5% threshold.
Arm/Group | GSK1562902A 18-60 YOA Group | GSK1562902A >60 YOA Group | Fluarix+Placebo 18-60 YOA Group | Fluarix+Placebo >60 YOA Group
Serious Adverse Events (participants affected / at risk) | 27/3397 | 15/405 | 10/1136 | 5/133
Other Adverse Events (participants affected / at risk) | 3189/3397 | 338/405 | 938/1136 | 83/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1562902A 18-60 YOA Group (N=3397) | GSK1562902A >60 YOA Group (N=405) | Fluarix+Placebo 18-60 YOA Group (N=1136) | Fluarix+Placebo >60 YOA Group (N=133)
Angina pectoris (Cardiac disorders) | 1 | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 2 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac valve (Cardiac disorders) | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 1
Macular hole (Eye disorders) | 0 | 0 | 0 | 1
Anal fissure (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oesophageal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0 | 0
Anaphylactic shock (Immune system disorders) | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Groin abscess (Infections and infestations) | 1 | 0 | 0 | 0
Mediastinitis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Genital injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Heat stroke (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Ligament injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Diabetes mellitus noninsulindependent (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Vitamin b12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Intra-uterine death (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Generalised anxiety disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0 | 0
Bartholinís cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Endometriosis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Varicose vein (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1562902A 18-60 YOA Group (N=3397) | GSK1562902A >60 YOA Group (N=405) | Fluarix+Placebo 18-60 YOA Group (N=1136) | Fluarix+Placebo >60 YOA Group (N=133)
Ecchymosis (General disorders) | 320 | 29 | 65 | 5
Induration (General disorders) | 1150 | 108 | 215 | 19
Pain (General disorders) | 3037 | 271 | 748 | 39
Redness (General disorders) | 1277 | 165 | 312 | 38
Swelling (General disorders) | 1107 | 133 | 196 | 17
Arthralgia (General disorders) | 874 | 82 | 130 | 15
Fatigue (General disorders) | 1736 | 117 | 346 | 24
Fever (General disorders) | 466 | 24 | 38 | 9
Headache (General disorders) | 1566 | 114 | 350 | 19
Myalgia (General disorders) | 1670 | 124 | 276 | 18
Shivering (General disorders) | 711 | 26 | 86 | 5
Sweating (General disorders) | 727 | 64 | 134 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.